CLINICAL TRIAL: NCT02935517
Title: A Multiple-Site, Phase 1/2, Safety and Efficacy Trial of AGTC 402, a Recombinant Adeno-associated Virus Vector Expressing CNGA3, in Patients With Congenital Achromatopsia Caused by Mutations in the CNGA3 Gene
Brief Title: Safety and Efficacy Trial of AAV Gene Therapy in Patients With CNGA3 Achromatopsia (A Clarity Clinical Trial)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beacon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGTC-CNGA3-002
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Achromatopsia
Keywords: Color vision deficiency; Color vision defects; Vision disorders; Sensation disorders; Neurologic manifestations; Nervous system diseases; Eye diseases; Signs and symptoms
MeSH Terms: conditions — Color Vision Defects; Vision Disorders; Sensation Disorders; Neurologic Manifestations; Nervous System Diseases; Eye Diseases; Signs and Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Group 1: 4.0 x 10^10 vg/mL of AGTC-402 (Experimental): Subjects at least 18 y/o treated with 4.0 x 10^10 vg/mL of rAAV2tYF-PR1/7-hCNGA3 study drug.
  Interventions: Biological: AGTC-402
- Group 2: 1.2 x 10^11 vg/mL of AGTC-402 (Experimental): Subjects at least 18 y/o treated with 1.2 x 10^11 vg/mL of rAAV2tYF-PR1/7-hCNGA3 study drug.
  Interventions: Biological: AGTC-402
- Group 3: 3.6 x 10^11 vg/mL of AGTC-402 (Experimental): Subjects at least 18 y/o treated with 3.6 x 10^11 vg/mL of rAAV2tYF-PR1/7-hCNGA3 study drug.
  Interventions: Biological: AGTC-402
- Group 3a: 3.6 x 10^11 vg/mL of AGTC-402 (Experimental): Subjects 6 to 17 y/o treated with 3.6 x 10^11 vg/mL of rAAV2tYF-PR1/7-hCNGA3 study drug.
  Interventions: Biological: AGTC-402
- Group 4: 1.1 x 10^12 vg/mL of AGTC-402 (Experimental): Subjects at least 18 y/o treated with 1.1 x 10^12 vg/mL of rAAV2tYF-PR1/7-hCNGA3 study drug.
  Interventions: Biological: AGTC-402
- Group 4a: 1.1 x 10^12 vg/mL of AGTC-402 (Experimental): Subjects 4 to 8 y/o treated with 1.1 x 10^12 vg/mL of rAAV2tYF-PR1/7-hCNGA3 study drug.
  Interventions: Biological: AGTC-402
- Group 5: 3.2 x 10^12 vg/mL of AGTC-402 (Experimental): Subjects at least 18 y/o treated with 3.2 x 10^12 vg/mL of rAAV2tYF-PR1/7-hCNGA3 study drug.
  Interventions: Biological: AGTC-402
- Group 6: MTD of AGTC-402 (Experimental): Subjects 4 to 8 y/o treated with a maximum tolerated dose of rAAV2tYF-PR1/7-hCNGA3 study drug determined by Groups 1-5.
  Interventions: Biological: AGTC-402

INTERVENTIONS:
Biological: AGTC-402 — AGTC-402 is a non-replicating, rep/cap-deleted, recombinant adeno-associated virus vector that expresses the CNGA3 gene.
  Other Names: rAAV2tYF-PR1.7-hCNGA3

SUMMARY:
This will be a non-randomized, open-label, Phase 1/2 study of the safety and efficacy of AGTC-402, administered to one eye by subretinal injection in individuals with achromatopsia caused by mutations in the CNGA3 gene. The primary study endpoint will be safety and the secondary study endpoint will be efficacy.

DETAILED DESCRIPTION:
This will be a non-randomized, open-label, Phase 1/2 study of the safety and efficacy of AGTC-402 administered to one eye by subretinal injection in individuals with achromatopsia caused by mutations in the CNGA3 gene. The primary study endpoint will be safety and the secondary study endpoint will be efficacy.

Subjects will be enrolled sequentially in six groups. Subjects in Groups 1, 2, 3, 4, and 5 will be at least 18 years of age and will receive varying dose levels of study agent. Subjects in Group 3a will be 6 to 17 years of age and will receive the same dose as Group 3. Subjects in Group 4a and 6 will be between 4 and 8 years of age. Subjects in Group 4a will receive the same dose as Group 4, and subjects in Group 6 will receive the maximum tolerated dose identified in Groups 1, 2, 3, 3a, 4, 4a, and 5.

Safety will be monitored by evaluation of ocular and non-ocular adverse events and hematology and clinical chemistry parameters. Efficacy parameters will include visual acuity, light discomfort testing, color vision, static visual field, ERG, adaptive optics retinal imaging, functional MRI (fMRI), color brightness test and OCT.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with documented mutations in both alleles of the CNGA3 gene;
2. Retinal disease consistent with a clinical diagnosis of achromatopsia;
3. At least 18 years of age for Groups 1, 2, 3, 4, and 5. At least 6 years of age for Group 3a, and and 4-8 years of age for Groups 4a and 6;
4. Able to perform tests of visual and retinal function;
5. Visual acuity in the study eye not better than 55 ETDRS letters (Snellen equivalent 20/80) based on the average of two examinations at the baseline visit;
6. Acceptable laboratory parameters;
7. For females of childbearing potential: A negative pregnancy test within 2 days before administration of study agent.

Exclusion Criteria include:

1. Best-corrected visual acuity difference between the two eyes of > 15 ETDRS letters (3 lines);
2. Evidence of degenerative myopia in the study eye;
3. Pre-existing eye conditions that would contribute to vision loss in either eye or increase the risk of subretinal injection in the study eye.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 1 year
  Proportion of participants experiencing grade 3 or greater adverse events

SECONDARY OUTCOMES:
Visual acuity | 1 year
  Changes in best corrected visual acuity compared to pre-treatment
Light aversion | 1 year
  Changes in light discomfort testing compared to pre-treatment
Color vision | 1 year
  Changes in color vision testing compared to pre-treatment

CONTACTS AND LOCATIONS:
Overall Officials: David Jacobs, MD, MBA, Study Director — Applied Genetics Technologies Corporation
Locations (6):
- United States (5):
  - VitreoRetinal Associates, Gainesville, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Casey Eye Institute, Oregon Health and Sciences University, Portland, Oregon
- Hadassah-Hebrew University Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banin E, Gootwine E, Obolensky A, Ezra-Elia R, Ejzenberg A, Zelinger L, Honig H, Rosov A, Yamin E, Sharon D, Averbukh E, Hauswirth WW, Ofri R. Gene Augmentation Therapy Restores Retinal Function and Visual Behavior in a Sheep Model of CNGA3 Achromatopsia. Mol Ther. 2015 Sep;23(9):1423-33. doi: 10.1038/mt.2015.114. Epub 2015 Jun 19. PMID 26087757
- See also: AGTC website — http://www.agtc.com